CLINICAL TRIAL: NCT00795132
Title: Reduced Intensity Conditioning Hematopoietic Cell Transplantation for Pediatric Patients With Hematologic Malignancies at High Risk for Transplant Related Mortality With Standard Transplantation
Brief Title: Hematopoietic Cell Transplantation for Pediatric Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI12073
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Acute Leukaemia; Chronic Disease; Leukemia; Myelodysplasia; Lymphoma
Keywords: cancer; Hematologic Malignancies; Hematopoietic Cell Transplantation
MeSH Terms: conditions — Chronic Disease; Leukemia; Anemia, Refractory, with Excess of Blasts; Lymphoma; Neoplasms; Hematologic Neoplasms | interventions — Busulfan; Antilymphocyte Serum; thymoglobulin; fludarabine; fludarabine phosphate; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Related BM PBSC (Active Comparator): Bone Marrow Peripheral Blood Stem Cell (BM PBSC) from a donor related to the participant/recipient
  Interventions: Drug: Busulfan; Drug: Anti-Thymocyte Globulin; Drug: Fludarabine; Drug: Cyclosporine; Drug: Mycophenolate mofetil
- Unrelated BM PBSC (Active Comparator): Bone Marrow Peripheral Blood Stem Cell (BM PBSC) from a donor unrelated to the participant/recipient
  Interventions: Drug: Busulfan; Drug: Anti-Thymocyte Globulin; Drug: Fludarabine; Drug: Cyclosporine; Drug: Mycophenolate mofetil
- Unrelated Blood Cord (Active Comparator): Blood Cord donated from a donor unrelated to the participant/recipient
  Interventions: Drug: Busulfan; Drug: Anti-Thymocyte Globulin; Drug: Fludarabine; Drug: Cyclosporine; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Busulfan — This drug is a bifunctional alkylating agent. Busulfan is highly toxic to noncycling or slowly-cycling cells. Pharmacokinetic studies of the IV formulation in pediatrics have shown that using a dose of 0.8mg/kg IV q6 hours most patients will achieve AUC levels between 800 and 1300 uM/min, representing steady state levels between 600-900ug/ml. The manufacturer recommends higher doses, 1.1mg/kg for children less than 12kg. Because this is a reduced intensity study and infants on the study will be very heavily pretreated we will use the lower dose of 0.8mg/kg q6 hours for a total of 8 doses for all patients.
  Other Names: Busulfex
Drug: Anti-Thymocyte Globulin — Thymoglobulin will be administered at a dose of 2.5 mg/kg recipient body weight intravenously on each of 4 successive mornings (Days -4, -3,-2,-1) for patients receiving unrelated grafts and at a dose of 2.5mg/kg as a single dose on d-1 for patients receiving related marrow grafts. ATG is infused over a minimum of 4 hours, but is generally better tolerated over 6-8 hours. Suggested premedications are acetaminophen (10 mg/kg/dose), diphenhydramine (1 mg/kg/dose), and methylprednisolone. The methylprednisolone should be given at a dose of
  1mg/kg 30 minutes prior to the ATG, with another 1mg /kg four hours into the infusion (total 2mg/kg/d). Patients are observed continuously for possible allergic reactions throughout the infusion.
  Other Names: Thymoglobulin® [Anti-thymocyte Globulin; (Rabbit)]
Drug: Fludarabine — Administration and Dosage: Fludarabine will be administered at a dose of 30 mg/m2 in 100 ml of D5W intravenously over one hour on each of six consecutive days -10 through -5 for unrelated grafts or d-7 through d-2 for related grafts. Fludarabine is a fluorinated nucleotide analog of the antiviral agent vidarabine, 9-beta-D-arabinofuranosyladenine. Fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoro-ara-ATP. The half-life of 2-fluoro-ara-A is approximately 10 hours. The mean total plasma clearance is 8.9 L/hr/m2 and the mean volume of distribution is 98 L/m2. Approximately 23% is excreted unchanged. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis.
  Other Names: Fludara
Drug: Cyclosporine — Cyclosporine is a potent immunosuppressive agent that in animals prolongs survival of allogeneic transplants involving skin, kidney, liver, heart, pancreas, bone marrow, small intestine, and lung. The effectiveness of cyclosporine results from specific and reversible inhibition of immunocompetent lymphocytes in the G 0 - and G
  1 -phase of the cell cycle. Administration and Dosage: Cyclosporin start on day -3 initially at a dose of 2.5mg/kg IV q12 hours or 3mg/kg/dose (neoral equivalent) PO q12 hours targeting suggested troughs of 250 to 350 ng/ml. Continuous infusion cyclosporin may be allowed per institutional preference. 3x daily dosing may be used for younger children to achieve therapeutic levels. PBMTC Protocol #ONC0313 19 Continuous infusion cyclosporin may be allowed per institutional preference.
Drug: Mycophenolate mofetil — MMF is a potent, selective, uncompetitive, and reversible inhibitor of inosine monophosphate dehydrogenase (IMPDH), and therefore inhibits the de novo pathway of guanosine nucleotide synthesis without incorporation into DNA. Administration and Dosage: Initial dosage will be IV or PO with switch to PO when tolerated. Starting doses will be 15 mg/kg/day bid (total dose 30mg/kg/d, IV same as PO dose) beginning day 0 with the first dose given approximately 4-6 hours after the stem cell infusion. This dose will stop on day +30 for patients receiving matched sibling BM/PBSC and UCB grafts, but will continue until day +40 and then taper at approximately 11%/wk over 8 weeks until patients are off at day +96.
  Other Names: MMF, CellCept

SUMMARY:
This is a phase II trial of reduced intensity conditioning with Bu/Flu/ATG in pediatric patients with hematologic malignancies at high risk for transplant related mortality with standard transplantation. Patients qualify based on organ system dysfunction, active but stable infection, history of previous transplant or late stage disease. We plan to enroll 45 patients through the Pediatric Blood and Marrow Transplant Consortium (PBMTC) and anticipate that the outcome of the trial will pave the way for phase II or III disease specific protocols addressing efficacy of the approach compared to standard transplant approaches in better risk patients.

DETAILED DESCRIPTION:
Summary/Proposal: Reduced Intensity Hematopoietic Cell Transplantation for High-Risk Relapsed Pediatric Hematologic Malignancies and Patients Ineligible for Standard Transplantation We propose a phase II trial of reduced intensity conditioning with Bu/Flu/ATG in pediatric patients with hematologic malignancies at high risk for transplant related mortality with standard transplantation. Patients qualify based on organ system dysfunction, active but stable infection, history of previous transplant, or late stage disease. We plan to enroll 45 patients through the Pediatric Blood and Marrow transplant Consortium (PBMTC) and anticipate that the outcome of the trial will pave the way for phase II or III disease specific protocols addressing efficacy of the approach compared to standard transplant approaches in better risk patients.

Hypothesis High risk pediatric hematologic malignancy patients ineligible for standard myeloablative HCT undergoing reduced intensity conditioning (RIC) HCT can achieve a sustained engraftment rate > 90% with a 100day TRM < 30% using either bone marrow or PBSC from related or unrelated donors. High risk pediatric patients undergoing RIC-HCT using related or unrelated cord blood can achieve a sustained engraftment rate >80% and a 100d TRM <30%.

Rationale for Reduced Intensity Approaches in High Risk Patients There are a number patient-specific risk factors associated with increased transplant related mortality. They can be broadly placed into three categories: pretransplant organ system dysfunction, active infections at the time of transplant, and degree of pretransplant therapy (previous transplants, third or subsequent remission, etc.).

The primary objective of this study is to determine the likelihood of achieving sustained donor engraftment using reduced intensity conditioning (fludarabine/busulfan/ATG) followed by hematopoietic cell transplantation (HCT) with either cord blood, bone marrow or peripheral blood stem cells (PBMTC) in pediatric patients with hematopoietic malignancies who are at high risk of transplant related mortality (TRM) with myeloablative HCT. Patients qualify based on organ system dysfunction, active but stable infection, history of previous transplant or late stage disease. We plan to enroll 45 patients through the Pediatric Blood and Marrow Transplant Consortium (PBMTC) and anticipate that the outcome of the trial will pave the way for phase II or III disease specific protocols addressing efficacy of the approach compared to standard transplant approaches in better risk patients.

Study procedures Patients receive their conditioning regimen consisting of fludarabine, busulfan, and ATG and then receive their stem cell transplant. Patients receive immunosuppression consisting of cyclosporine and mycophenolate mofetil. Patients with persistent or progressive disease may receive donor lymphocyte infusion off protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be age 21 or younger and must have hematologic malignancies treatable with allogeneic hematopoietic transplantation (acute and chronic leukemias, myelodysplasia or lymphomas, see protocol for further details). Patients qualify for this approach in four ways: 1) presence of organ system dysfunction or severe systemic infections that significantly increase transplant related mortality with standard myeloablative transplant regimens, 2) history of previous myeloablative allogeneic or autologous transplantation, 3) currently in a third or higher CR receiving an unrelated stem cell transplant, or 4) a combination of toxicities that leads the investigator to feel that the child is at high risk (>50%) of TRM. Patients eligible for inclusion based on consideration number 4 above cannot be enrolled unless discussed with the study chair.
2. Organ system dysfunction: at least one of the following organ system dysfunction criteria plus minimum organ function listed in exclusion criteria qualify a patient for treatment on this protocol

   1. Pulmonary: DLCO, FEV1 or TLC/FVC <60% predicted. Patients too young for PFTs with suspected pulmonary toxicity should be assessed by a consulting pulmonologist. If the pulmonologist judges the child to have moderate-severe pulmonary disease they qualify for inclusion.
   2. Renal: creatinine clearance <60ml/m/1.73m2
   3. Hepatic: transaminases >4x normal or total bilirubin >2.0
   4. Cardiac: all patients with suspected cardiac toxicity should undergo a cardiac echo. If the shortening fraction (SF) is <25% a measurement of ejection fraction must be obtained. Patients qualify for reduced intensity therapy if the SF is <25% and the EF <50%.
3. Infections: Patients with responsive but unresolved invasive infections. These infections may be fungal, bacterial or other opportunistic infections. Viral infections do not meet this eligibility criteria.
4. Other patient groups at high risk for transplant related mortality: Patients with a history of a prior allogeneic or autologous transplantation and patients who are in CR3 or greater and receiving an unrelated stem cell transplant are also eligible for this protocol. If the investigator feels that a patient has a combination of risk factors that could increase their risk of transplant related mortality to >50% with standard transplantation they may be eligible for inclusion, but such patients must be reviewed with the protocol chairman prior to enrollment.

Exclusion Criteria:

1. Patients must be in a CR (<5% blasts on BM morphology, no active CNS disease, see protocol) with the following exceptions:

   1. AML may proceed with M2 marrow status (<20% blasts).
   2. Lymphoma: residual disease must be responsive and non-bulky (<5cm largest diameter).
   3. Myelodysplasia: Patients with RA, and RAEB are eligible, but RAEB-IT patients are only eligible if treated to <5% blasts (RA) with chemotherapy.
   4. CML-BP must be treated to CR/CP2 to be eligible.
2. Females who are pregnant
3. Patients who are HIV positive or who have other progressive infections
4. Organ dysfunction: patients are ineligible for the following levels of severe organ system dysfunction:

   1. Cardiac: Ejection fraction <30%
   2. Pulmonary: Receiving continuous supplementary oxygen or any of the following: DLCO <30%, FVC/TLC < 30% or FEV1 <30%
   3. Hepatic: patients will be excluded for hepatic synthetic dysfunction evidenced by any of the following: prolongation of the prothrombin time with an INR >2.0, total serum bilirubin >3, or transaminases >10x normal.
   4. Renal: patients with a creatinine clearance <30ml/m/1.73m2 or who require dialysis are not eligible

Donor Eligibility Criteria:

1. Related or unrelated donor who is a 6/6 HLA match at HLA-A, B, and DRB1 locus. 5/6 matches are acceptable with mismatches at class I alleles (A and B), but DRB1 mismatches are not allowed. Intermediate resolution typing of class I and high resolution typing of class II alleles is required. (HLA-C and HLA-DQ matching is encouraged, but not required with the ideal donor matching at 10/10 alleles.)
2. Unrelated cord blood may be used if matched at HLA-A, B and DRB1 at either 4/6, 5/6, or 6/6 antigens. The minimum mononuclear cell dose required for eligibility is 3 x 107 mononuclear cells/kg recipient body weight (based on frozen cell dose). It is strongly suggested that a back up unit of umbilical cord blood be reserved, though not requested, in case of rejection.

Donors must pass required institutional and NMDP health and infectious disease screening.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2004-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Principal Investigator — Primary Children's Hospital
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Pulsipher MA, Boucher KM, Wall D, Frangoul H, Duval M, Goyal RK, Shaw PJ, Haight AE, Grimley M, Grupp SA, Kletzel M, Kadota R. Reduced-intensity allogeneic transplantation in pediatric patients ineligible for myeloablative therapy: results of the Pediatric Blood and Marrow Transplant Consortium Study ONC0313. Blood. 2009 Aug 13;114(7):1429-36. doi: 10.1182/blood-2009-01-196303. Epub 2009 Jun 15. PMID 19528536

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: This group contains data from all groups (Related Bone marrow Peripheral Blood Stem Cell (BM PBSC), Unrelated Peripheral Blood Stem Cell (PBSC), and Unrelated Cord blood.
Period: Overall Study
Arm/Group | All Study Participants
Started | 47
Completed | 44
Not Completed | 3
Not completed — Death | 1
Not completed — Relapse | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13 (9.899)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 35
  Canada | 8
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of High Risk Pediatric Patients With Successful Sustained Donor Engraftments
Description: Assessed donor engraftment in very high risk pediatric patients.
Time Frame: 24 months
Population: All enrolled patients were analyzed except for the 3 patients who relapsed or died prior to engraftment.
Measure: Number; unit: participants
Groups:
- Related BM PBSC: Related donor: bone marrow or peripheral blood stem cell (PBSC)
- Unrelated BM PBSC: Unrelated donor: bone marrow or peripheral blood stem cell (PBSC)
- Unrelated Cord Blood: Unrelated donor: Cord Blood
Arm/Group | Related BM PBSC | Unrelated BM PBSC | Unrelated Cord Blood
Number analyzed (Participants) | 16 | 18 | 10
participants | 16 | 18 | 10

2. Secondary Outcome: Two Year Overall Survival
Description: The probability that a given patient will be alive two years after transplantation.
Time Frame: 24 months
Population: All enrolled participants were analyzed.
Measure: Mean (Standard Error); unit: probability
Groups:
- Related BM PBSC; Unrelated BM PBSC; Unrelated Cord Blood: All participants were analyzed.
Arm/Group | Related BM PBSC | Unrelated BM PBSC | Unrelated Cord Blood
Number analyzed (Participants) | 16 | 19 | 12
probability | 0.501 (0.141) | 0.395 (0.120) | 0.438 (0.165)

3. Secondary Outcome: Number of Participants Who Experienced Transplantation-related Mortality (TRM)
Description: Cumulative incidence transplantation-related mortality (TRM)
Time Frame: 24 months
Population: All incidences of enrolled patients were analyzed.
Measure: Number; unit: participants
Groups:
- Related BM PBSC; Unrelated BM PBSC; Unrelated Cord Blood: All incidences of enrolled patients were analyzed.
Arm/Group | Related BM PBSC | Unrelated BM PBSC | Unrelated Cord Blood
Number analyzed (Participants) | 16 | 19 | 12
participants | 0 | 5 | 1

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

LIMITATIONS AND CAVEATS:
Participants who experienced early relapse or death before engraftment were excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes